CLINICAL TRIAL: NCT02528799
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Tolerability of Nexvax2 Preceded by a Dose Titration Period in Subjects With Celiac Disease Currently on a Gluten-Free Diet
Brief Title: Safety and Tolerability of Nexvax2 in Subjects With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmusanT, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nexvax2-1004; U1111-1173-7522 (Other: New Zealand Universal Trial Number (UTN))
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2017-04

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease | interventions — Nexvax2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Nexvax2 DQ2.5 Homozygotes (Cohort 1) (Experimental): Nexvax2 by ID injections for a total of 14 doses over 46 days.
  Interventions: Biological: Nexvax2
- Nexvax2 Placebo DQ2.5 Homozygotes (Cohort 1) (Placebo Comparator): Nexvax2 Placebo by ID injections for a total of 14 doses over 46 days.
  Interventions: Biological: Nexvax2 placebo
- Nexvax2 DQ2.5 Non-homozygotes (Cohort 2) (Experimental): Nexvax2 by ID injections for a total of 14 doses over 46 days.
  Interventions: Biological: Nexvax2
- Nexvax2 Placebo DQ2.5 Non-homozygotes (Cohort 2) (Placebo Comparator): Nexvax2 Placebo by ID injections for a total of 14 doses over 46 days.
  Interventions: Biological: Nexvax2 placebo
- Nexvax2 DQ2.5 Non-homozygotes (Cohort 3) (Experimental): Nexvax2 by ID injections for 18 doses (up to 27 doses) over 60 days (maximum of 91 days).
  Interventions: Biological: Nexvax2
- Nexvax2 Placebo DQ2.5 Non-homozygotes (Cohort 3) (Placebo Comparator): Nexvax2 Placebo by ID injections for 18 doses (up to 27 doses) over 60 days (maximum of 91 days).
  Interventions: Biological: Nexvax2 placebo

INTERVENTIONS:
Biological: Nexvax2 — Nexvax2 intra-dermal injections twice weekly
  Arms: Nexvax2 DQ2.5 Homozygotes (Cohort 1); Nexvax2 DQ2.5 Non-homozygotes (Cohort 2); Nexvax2 DQ2.5 Non-homozygotes (Cohort 3)
Biological: Nexvax2 placebo — Sodium chloride 0.9% intra-dermal injections twice weekly
  Arms: Nexvax2 Placebo DQ2.5 Homozygotes (Cohort 1); Nexvax2 Placebo DQ2.5 Non-homozygotes (Cohort 2); Nexvax2 Placebo DQ2.5 Non-homozygotes (Cohort 3)

SUMMARY:
A randomized, double-blind, placebo-controlled, dose titration trial, stratified by Human Leukocyte Antigen (HLA)-DQ2.5 genotype in subjects with celiac disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, study to evaluate the safety and tolerability of Nexvax2 preceded by dose titration period in patients with celiac disease currently on a gluten-free diet. The study will consist of a Screening Period, a Treatment Period, and a Follow-up Period. Eligible subjects will be enrolled in one of three cohorts according to whether they are homozygous or not homozygous for both genes coding for HLA-DQ2.5.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and understands the informed consent form before initiation of any study specific procedures.
2. Subject is between 18 and 70 years old (inclusive) on the date of the Screening Visit.
3. Subject has been diagnosed with celiac disease on the basis of intestinal histology showing villous atrophy according to expert guidelines current at the time of diagnosis.
4. Subject has HLA DQ2.5 genotype (HLA-DQA1*05 and HLA-DQB1*02).

Exclusion Criteria:

1. Subject has not been maintained on a gluten-free diet for at least 1 year.
2. Celiac Dietary Adherence Test at screening indicates non-compliance to gluten-free diet (score >12).
3. Serum levels of both recombinant human transglutaminase (tTG)-specific immunoglobulin-A (IgA) and deamidated gliadin peptide (DGP)-specific immunoglobulin-G (IgG) are elevated above the manufacturer's upper limit of normal. The elevation of one or other of the serology test for tTG IgA and DGP IgG is not an exclusion.
4. Subject has uncontrolled complications of celiac disease or a medical condition which, in the opinion of the investigator, would impact the immune response or pose an increased risk to the subject.
5. Subject is or has been using an immuno-modulatory or immune suppressing medical treatment during the 2 months prior to Screening, for example azathioprine, methotrexate, or biological
6. Subject is female and premenopausal or perimenopausal and has a male partner who is not sterile, unless she is sterile, or she practices true abstinence, or unless throughout the entire study period and for 30 days after study drug discontinuation she is using a medically acceptable method of contraception.
7. Subject is male with a premenopausal or perimenopausal female partner who is not sterile, unless he is sterile, or he practices true abstinence, or unless throughout the entire study period and for 30 days after study drug discontinuation he is using a medically acceptable method of contraception, or unless his female partner is using a medically acceptable method of contraception.
8. Subject is unable and/or unwilling to comply with study requirements.
9. Subject has taken oral or parenteral corticosteroids within the previous six weeks prior to Screening. Topical or inhaled corticosteroids are acceptable.
10. Subject has received an experimental therapy within 30 days prior to Screening.
11. Subject has previously been enrolled and dosed in a clinical trial with Nevax2.
12. Subject has any of the following laboratory abnormalities at Screening:

    * Alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) ≥ 2 × the upper limit of normal (ULN)
    * Hemoglobin <10 g/dL
    * Platelet count <100 × 109/L
    * White blood cell count (WBC) outside the normal range and judged clinically significant by the investigator
    * Direct bilirubin outside the normal range
    * Any other clinically significant abnormal laboratory values, as determined by the investigator
13. Subject is lactating, is known to be pregnant, has a positive pregnancy test at Screening or Treatment Day, intends to become pregnant, or is nursing.
14. Subject has a history or presence of any medically significant condition considered by the investigator to have the potential to adversely affect participation in the study and/or interpretation of the study results.
15. Subject has a history of severe allergic reactions (e.g., swelling of the mouth and throat, difficulty breathing, hypotension, or shock) that require medical intervention.
16. Subject has donated blood ≤ 56 days prior to Screening and plans to donate blood within 5 weeks after study completion.
17. Subject has a clinically relevant abnormality on electrocardiogram (ECG), as determined by the investigator.
18. Other unspecified reasons that in the opinion of the investigator or the sponsor make the subject unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-08; Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity and safety of Nexvax2 according to the "Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0" | Treatment Period (~7 to 9 weeks)
  Number and Percentage of Participants with Treatment-related Adverse Events assessed by the "Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 will be tabulated using counts and proportions detailing frequently occurring, serious and severe events. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to study treatments.

SECONDARY OUTCOMES:
Weekly Gastrointestinal Symptom Rating Scale (GSRS) | Treatment Period (~7 to 9 weeks)
  The GSRS score is the average weekly scores for 15 symptoms rated on a 7-point severity scale. GSRS scores over the 6-week Treatment Period will be compared.
Plasma Cytokine Levels | Treatment Period (~7 to 9 weeks)
  The relative change from pre-dose levels up to 10 hours after dosing in the concentration of plasma cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Robert P. Anderson, MB ChB, PhD, Study Chair — ImmusanT, Inc.
Locations (4):
- Australia (3):
  - Q-Pharm Pty Ltd., Herston, Queensland
  - CMAX, A Division of IDT Australia Ltd, Adelaide, South Australia
  - Linear Clinical Research, Nedlands
- Auckland Clinical Studies Ltd, Auckland, New Zealand

REFERENCES:
- [Derived] Daveson AJM, Ee HC, Andrews JM, King T, Goldstein KE, Dzuris JL, MacDougall JA, Williams LJ, Treohan A, Cooreman MP, Anderson RP. Epitope-Specific Immunotherapy Targeting CD4-Positive T Cells in Celiac Disease: Safety, Pharmacokinetics, and Effects on Intestinal Histology and Plasma Cytokines with Escalating Dose Regimens of Nexvax2 in a Randomized, Double-Blind, Placebo-Controlled Phase 1 Study. EBioMedicine. 2017 Dec;26:78-90. doi: 10.1016/j.ebiom.2017.11.018. Epub 2017 Nov 22. PMID 29191561
- See also: MedlinePlus — http://www.nlm.nih.gov/medlineplus/
- See also: ImmusanT, Inc. — http://www.immusant.com/